CLINICAL TRIAL: NCT01244373
Title: Observational Case Series of the Implantation of Intraocular Lens "QUATRIX® Aspheric Evolutive Pre-loaded".
Brief Title: A Prospective Observational Case Series of a Four-ring-haptic Acrylic One-piece IOL
Acronym: Qu01
Status: Completed | Type: Observational
Sponsor: General Hospital Linz (Other)
Collaborators: Department of ophthalmology, General Hospital Linz (Unknown)
Responsible Party: PD Dr. Siegfried G. Priglinger
Other Study IDs: Quatrix01
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Cataract
Keywords: Best-corrected visual acuity; posterior capsule opacification; QUATRIX® Aspheric Evolutive pre-loaded
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with senile cataract: Patients with senile cataract

SUMMARY:
To describe biocompatibility, postoperative results and complications after implantation of the Corneal Quatrix Evolutive (Corneal, Croma, Austria) intraocular lens, a hydrophilic acrylic intraocular lens (IOL) with 4-haptic design and 360° sharp optic edge.

DETAILED DESCRIPTION:
In this prospective case series the Corneal Quatrix Evolutive IOL was implanted in 14 eyes of nine patients with senile cortico-nuclear cataract. A standardized surgical technique and post-operative regimen were applied. Six months postoperatively best corrected visual acuity (BCVA), refraction and complications (especially) posterior capsule opacification (PCO) were analysed.

ELIGIBILITY:
Inclusion Criteria:

Patients with senile cortico-nuclear cataracts without previous intraocular surgery

Exclusion Criteria:

* Dilated pupil size of < 6 mm
* long-term anti-inflammatory treatment
* previous history of intraocular surgery
* previous history of corneal endothelial damage
* previous history of ocular trauma
* traumatic cataract
* history of uveitis
* diabetic retinopathy
* advanced macular degeneration

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced age-related cataract and indication for phacoemuslification of the lens with following implantation of an intraocular lens (posterior chamber)
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2008-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Best-corrected visual acuity (BCVA) | Six months
  The best-corrected visual acuity is assessed with glasses after cataract operation

SECONDARY OUTCOMES:
Posterior capsule opacification | Six months
  The posterior capsule opacification is assessed by slit lamp examination and subjective grading

CONTACTS AND LOCATIONS:
Locations (1):
- Department of ophthalmology, General Hospital Linz, Linz, Upper Austria, Austria

REFERENCES:
- [Background] Kramer S, Schroder AC, Bruckner K, Jonescu-Cuypers C, Seitz B. [Subluxation of hydrophilic acrylate intraocular lenses due to massive capsular fibrosis]. Ophthalmologe. 2010 May;107(5):460-4. doi: 10.1007/s00347-009-2025-y. German. PMID 19756637
- [Background] Michael K, O'Colmain U, Vallance JH, Cormack TG. Capsule contraction syndrome with haptic deformation and flexion. J Cataract Refract Surg. 2010 Apr;36(4):686-9. doi: 10.1016/j.jcrs.2009.09.042. PMID 20362866